CLINICAL TRIAL: NCT00829634
Title: Steady State Kinetics of l-Methamphetamine and Validation of Sensitivity of Dose Estimation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: San Francisco General Hospital (Other); University of California, San Francisco (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 27.092
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Nasal Congestion
Keywords: methamphetamine; inpatient; d-MA; l-MA; APRL; San Francisco; metabolism; Metabolism of methamphetamine
MeSH Terms: conditions — Nasal Obstruction | interventions — N-myristoyl-alaninol

ARMS (1):
- l-methamphetamine (Other)
  Interventions: Drug: l-methamphetamine; Drug: d-methamphetamine

INTERVENTIONS:
Drug: l-methamphetamine — 5mg of l-methamphetamine per day throughout the 2 week study
  Other Names: l-MA
Drug: d-methamphetamine — 15mg on Study Day 9, 30mg on Study Day 11, 45mg on Study Day 13
  Other Names: d-MA

SUMMARY:
The intent of this study is to see if the rate that the body breaks down l-methamphetamine (l-MA) could be used as an accurate estimate for the rate that the body breaks down d-methamphetamine (d-MA). l-MA is sold over the counter as a nasal decongestant where as d-MA is the commonly abused form of methamphetamine.

DETAILED DESCRIPTION:
Subjects will screen at St. Luke's Hospital in San Francisco to determine their eligibility.

Once enrolled the study will take two weeks. During the first week subjects attend daily, hour-long outpatient visits at San Francisco General Hospital. At these visits subjects will receive an oral dose of l-methamphetamine, have their vitals read, answer questionnaires and receive a blood draw.

During the second week of the study subjects are admitted to San Francisco General Hospital for a week long inpatient stay. During this stay the subject continues to receive l-methamphetamine but also receives three doses of d-methamphetamine on three separate days. In addition the subject receives blood draws, has their urine collected, and answers questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males and Females Between the Ages of 18 and 50
* Must have some experience with methamphetamine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Serum samples | Predose and Multiple Timepoints Post Doses
Urine Samples | 24 Hour Inpatient Collection

SECONDARY OUTCOMES:
Questionnaries | Predose and Multiple Timepoints Post Doses

CONTACTS AND LOCATIONS:
Locations (1):
- CPMC Addiction & Pharmacology Research Laboratory (APRL), San Francisco, California, United States